CLINICAL TRIAL: NCT03905642
Title: Multidose Safety and Tolerability Study of Dose Escalation of Liposomal Amikacin for Inhalation (ARIKAYCE™) in Cystic Fibrosis Patients With Chronic Infections Due to Pseudomonas Aeruginosa
Brief Title: Study of Dose Escalation of Liposomal Amikacin for Inhalation (ARIKAYCE™) - Extension Phase
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR02-105 Extension
Record Dates: First submitted 2019-04-02; First posted 2019-04-05 (Actual); Results first posted 2019-05-14 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Respiratory Infections; Pulmonary Cystic Fibrosis; CFTR
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Extension phase for evaluation of safety, tolerability and efficacy. Single dose group of 560 mg of Arikase TM
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 560 mg Arikayce™ (Experimental): Subjects in this cohort will receive 560 mg of Arikayce™
  Interventions: Drug: Arikayce™

INTERVENTIONS:
Drug: Arikayce™ — Amikacin (aminoglycoside) in a liposomal formulation.
  Other Names: Liposomal amikacin inhalation, LAI

SUMMARY:
A major factor in the respiratory health of cystic fibrosis (CF) patients is acquisition of chronic Pseudomonas (P.) aeruginosa infections. The infection rate with P. aeruginosa increases with age and by age 18 years, 80% of patients with CF in the U.S. are infected. Liposomal amikacin for inhalation (LAI; Arikayce™) is a sterile aqueous liposomal suspension consisting of amikacin sulfate encapsulated in liposomes. This formulation of amikacin maximizes the achievable dose and delivery to the lungs of infected patients when delivered via a nebulizer. Because liposome particles are small enough to penetrate and diffuse through sputum into the bacterial biofilm, they deposit drug close to the bacterial colonies (Meers, et al., 2008) (Clancy, et al., 2013), thus improving the bioavailability of amikacin at the infection site. The clinically achievable doses of amikacin in the LAI formulation can effectively increase the half-life of the drug in the lungs, and decrease the potential for systemic toxicity. LAI offers several advantages over current therapies in treating patients with CF with chronic infection caused by P. aeruginosa.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a genetic disease resulting from mutations in a 230 kb gene on chromosome 7 known as the cystic fibrosis transmembrane conductance regulator (CFTR). Patients with CF manifest pathological changes in a variety of organs that express CFTR. The lungs are frequently affected, the sequelae being chronic infections and airway inflammation. The principal goal of treatment of patients with CF is to slow the chronic deterioration of lung function.

This study is a Phase 2 study to evaluate the longer term safety, tolerability and efficacy of 560 mg once daily dose of Arikayce™ administered for 6 cycles over 18 months. Each cycle comprises 28 days of treatment followed by 56 days off treatment.

All study patients will receive study drug by inhalation via a PARI® eFlow nebulizer. All study patients will be followed for safety, pharmacokinetics (PK), clinical, and microbiologic activity for 28 days post completion of study treatment.

The original TR02-105 study was a Phase 2a study of safety and tolerability of 28 days of daily dosing of two dose cohorts (280 mg and 560 mg) of Arikayce™ versus placebo. Study subjects were randomized to receive either study drug or placebo (1.5% NaCl) by inhalation via a PARI® eFlow nebulizer. Cohort 1 (280 mg) completed 28 days of daily dosing with Arikayce™ and 14-day post-dosing safety evaluation by the Safety Committee before initiation of enrollment in Cohort 2 (560 mg). Cohort 2 completed 28 days of daily dosing, and a 14-day post-dosing safety assessment by the Data Safety and Monitoring Board (DSMB) to evaluate safety data. All study patients were followed for safety, PK and clinical and microbiologic activity for 28 days post completion of study treatment. Details of the original study are provided at ClinicalTrials.gov ID NCT00777296.

DSMB has recommended the amendment of the main study to evaluate safety and efficacy of additional cycles of treatment with Arikayce™. All patients who were randomized in the main study, were compliant with the study protocol, and continue meeting study eligibility criteria can be consented to participate in the open-label extension to evaluate the safety, tolerability, and efficacy of 560 mg once daily dose of Arikayce™ administered for 6 cycles over 18 months. Each cycle comprises 28 days of treatment followed by 56 days off treatment.

Clinical laboratory parameters, audiology testing, clinical adverse events and pulmonary function will be evaluated for all study subjects in order to determine the longer term safety, tolerability, and efficacy of Arikayce™. Serum specimens will be collected at periodic intervals to assess PK for safety. Additionally, sputum samples will be collected to determine changes in bacterial density. Pulmonary function testing and Cystic Fibrosis Questionnaire-Revised (CFQ-R) measurements will be assessed at selected time points throughout the study. Arikace™, Arikayce™, Liposomal Amikacin for Inhalation (LAI), and Amikacin Liposome Inhalation Suspension (ALIS) may be used interchangeably throughout this study and other studies evaluating amikacin liposome inhalation suspension.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient or designated legal guardian prior to the performance of any study related procedures.
2. Male or female study subjects ≥ 6 years of age or older.
3. Confirmed diagnosis of CF defined as a positive sweat chloride > 60 milliequivalents (mEq)/liter (by pilocarpine iontophoresis) and/or a genotype with 2 identifiable mutations consistent with CF accompanied by one or more clinical features of the CF phenotype.
4. History of chronic infection with P. aeruginosa (defined as 3 documented positive cultures in the prior 2 years of which at least one was obtained in the 3 months prior to randomization). The cultures could be obtained from the following respiratory secretions: sputum, throat swabs, nasopharyngeal swabs, or broncho-alveolar lavage fluid specimens.
5. Study subjects must produce a screening specimen (expectorated or induced sputum, throat swabs, nasopharyngeal swabs, or broncho-alveolar lavage fluid) that is positive for growth of P. aeruginosa.
6. FEV1 ≥ 40% of predicted at Screening.
7. SaO2 ≥ 90% at Screening while breathing room air.
8. Ability to comply with study medication use, study visits, and study procedures as judged by the investigator.
9. Ability to produce 0.5 grams sputum or be willing to undergo an induction to produce sputum for clinical evaluation.
10. Clinically stable with no evidence of acute upper or lower respiratory tract infection or history of pulmonary exacerbation within the 4 weeks prior to Screening.

Main criteria for inclusion of patients participating in the 18-month extension period:

1. Written informed consent obtained from the patient or designated legal guardian prior to the performance of any study-related procedures in the extension period.
2. Patient meets all of the above listed inclusion criteria (1-10) of the main protocol.

Exclusion Criteria:

1. Administration of any investigational drug within 8 weeks prior to Screening.
2. Emergency room visit or hospitalization for CF or respiratory-related illness within the 4 weeks prior to Screening.
3. History of alcohol, medication, or illicit drug abuse within the 1 year prior to Screening.
4. History of lung transplantation.
5. Female of childbearing potential who is lactating or is not practicing an acceptable method of birth control (e.g., abstinence, hormonal or barrier methods, partner sterilization, or IUD).
6. Positive pregnancy test. All women of childbearing potential will be tested.
7. Use of any anti-pseudomonal antibiotics (IV antibiotics, all inhalation antibiotics, oral fluoroquinolones) within the 28 days prior to Screening.
8. Initiation of chronic therapy (i.e. TOBI®, high-dose ibuprofen, rhDNase, macrolide antibiotics) within the 28 days prior to Screening.
9. History of sputum or throat swab culture yielding Burkholderia cepacia within 2 years of Screening.
10. History of mycobacterial and/or Aspergillus infection requiring treatment within 2 years prior to Screening, and/or history of allergic bronchopulmonary aspergillosis (ABPA).
11. History of biliary cirrhosis with portal hypertension, or splenomegaly (refer to study manual).
12. GGT, AST, or ALT ≥ 3 times the upper limit of normal at Screening visit.
13. ANC ≤ 1000 performed at Screening visit.
14. Serum creatinine > 1.5 times normal performed at Screening visit.
15. History of daily, continuous oxygen supplementation or requirement for more than 2 L/min at night.
16. Change in chest x-ray at Screening (or within the 3 months prior to Screening) with new onset infiltrates or that which compromise the safety of the study patient or the quality of the study data.

Main criteria for exclusion of patients participating in the 18 months extension period:

1. Patient meets any criteria for exclusion as listed above in the main protocol.
2. Patient who met any criteria for study drug discontinuation in the main protocol (TR02-105).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-01-08 (Actual); Primary Completion 2010-11-02 (Actual); Study Completion 2010-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Eagle, MD, Study Director — Insmed Incorporated
Locations (11):
- Leuven, Belgium
- Hungary (2):
  - Budapest
  - Kaposvár
- Skopje, North Macedonia
- Poland (2):
  - Rabka-Zdrój
  - Warsaw
- Belgrade, Serbia
- Slovakia (2):
  - Bratislava
  - Košice
- Ukraine (2):
  - Kharkiv
  - Kiev

REFERENCES:
- [Background] Clancy JP, Dupont L, Konstan MW, Billings J, Fustik S, Goss CH, Lymp J, Minic P, Quittner AL, Rubenstein RC, Young KR, Saiman L, Burns JL, Govan JR, Ramsey B, Gupta R; Arikace Study Group. Phase II studies of nebulised Arikace in CF patients with Pseudomonas aeruginosa infection. Thorax. 2013 Sep;68(9):818-25. doi: 10.1136/thoraxjnl-2012-202230. Epub 2013 Jun 8. PMID 23749840

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 560 mg Arikayce™
Started | 49
Completed | 41
Not Completed | 8
Not completed — Withdrawal by Subject | 3
Not completed — Pregnancy | 1
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Completed study but not 24 of 28 days | 2

BASELINE CHARACTERISTICS:
Arm/Group | 560 mg Arikayce™
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] — Age, 8-31 years
  years | 17.4 (6.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 20
FEV1 % predicted [Mean (Standard Deviation); unit: Percent %] | 59.73 (20.047)
P. aeruginosa density [Mean (Standard Deviation); unit: Log10 CFU/mL] — Population: Safety population
  Log10 CFU/mL
    number analyzed (Participants) | 44
    (all) | 6.289 (2.8587)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event Profile of 560 mg Once Daily Dose of Arikayce™ Administered for Six Cycles Over Eighteen Months.
Description: Number of Participants with indicated Adverse Events in subjects receiving 560 mg once daily dose of Arikayce™ administered for 6 cycles over 18 months.
Time Frame: 18 Months
Measure: Number; unit: participants
Arm/Group | 560 mg Arikayce™
Number analyzed (Participants) | 49
participants
  Any Adverse Event | 48
  Treatment-related adverse events | 15
  Grade 1: Mild | 28
  Grade 2: Moderate | 15
  Grade 3: Severe | 4
  Grade 4: Life-threatening or disabling | 1
  Grade 5: Death | 0
  Serious Adverse Events | 15
  Treatment-related serious adverse events | 0
  Deaths | 0
  Permanent discontinuations due to adverse events | 1

2. Secondary Outcome: FEV1 % Predicted
Description: A summary of relative change from extension study baseline time points in FEV1 % predicted is presented for the overall safety population and by treatment received.
Time Frame: Baseline, Days1, 14, 28, 56, 70, 85, 98, 112, 140, 154, 169, 182,196, 224, 238, 253, 266, 280, 308, 322, 337, 350, 364, 392, 406, 421, 434, 448, 476, 490, and 504
Population: Safety population
Measure: Mean (Standard Deviation); unit: Percent (%) predicted
Arm/Group | 560 mg Arikayce™
Number analyzed (Participants) | 49
Percent (%) predicted
  Baseline | 59.73 (20.047)
  Day 1: number analyzed (Participants) | 47
  Day 1 | 3.13 (8.553)
  Day 14: number analyzed (Participants) | 46
  Day 14 | 7.62 (15.246)
  Day 28: number analyzed (Participants) | 46
  Day 28 | 6.83 (14.593)
  Day 56: number analyzed (Participants) | 47
  Day 56 | 3.02 (11.174)
  Day 70: number analyzed (Participants) | 48
  Day 70 | 2.96 (13.580)
  Day 85: number analyzed (Participants) | 48
  Day 85 | 4.04 (15.450)
  Day 98: number analyzed (Participants) | 48
  Day 98 | 9.97 (16.594)
  Day 112: number analyzed (Participants) | 48
  Day 112 | 8.19 (20.116)
  Day 140: number analyzed (Participants) | 47
  Day 140 | 4.86 (19.337)
  Day 154: number analyzed (Participants) | 47
  Day 154 | 6.76 (20.633)
  Day 169: number analyzed (Participants) | 46
  Day 169 | 3.90 (19.141)
  Day 182: number analyzed (Participants) | 46
  Day 182 | 10.22 (18.349)
  Day 196: number analyzed (Participants) | 46
  Day 196 | 7.56 (20.607)
  Day 224: number analyzed (Participants) | 46
  Day 224 | 2.57 (19.165)
  Day 238: number analyzed (Participants) | 45
  Day 238 | 5.46 (17.872)
  Day 253: number analyzed (Participants) | 45
  Day 253 | 3.37 (17.755)
  Day 266: number analyzed (Participants) | 45
  Day 266 | 9.07 (19.747)
  Day 280: number analyzed (Participants) | 45
  Day 280 | 8.54 (19.179)
  Day 308: number analyzed (Participants) | 46
  Day 308 | 5.77 (19.633)
  Day 322: number analyzed (Participants) | 45
  Day 322 | 5.25 (20.946)
  Day 337: number analyzed (Participants) | 44
  Day 337 | 5.18 (21.740)
  Day 350: number analyzed (Participants) | 44
  Day 350 | 10.49 (21.615)
  Day 364: number analyzed (Participants) | 44
  Day 364 | 3.82 (18.895)
  Day 392: number analyzed (Participants) | 43
  Day 392 | 3.07 (18.380)
  Day 406: number analyzed (Participants) | 43
  Day 406 | 2.74 (18.301)
  Day 421: number analyzed (Participants) | 43
  Day 421 | 1.63 (19.094)
  Day 434: number analyzed (Participants) | 43
  Day 434 | 7.11 (20.022)
  Day 448: number analyzed (Participants) | 43
  Day 448 | 5.66 (20.422)
  Day 476: number analyzed (Participants) | 43
  Day 476 | 0.83 (21.741)
  Day 490: number analyzed (Participants) | 43
  Day 490 | 1.61 (19.922)
  Day 504: number analyzed (Participants) | 42
  Day 504 | 0.06 (22.196)

3. Secondary Outcome: Absolute Change in Sputum Density
Description: A summary of change from extension study baseline to all post-baseline time points during the treatment periods and at the end of the off-treatment periods in P aeruginosa sputum density (log10 CFU/mL) is presented for the overall safety population and by treatment received.
Time Frame: Baseline, Days 14, 28, 85, 98, 112, 140, 169, 182,196, 253, 266, 280, 337, 350, 364, 421, 434, and 448
Population: Per Protocol population defined as all patients who completed at least 24 of the 28 days of dosing for each of the 6 cycles
Measure: Mean (Standard Deviation); unit: Log 10 CFU/mL
Arm/Group | 560 mg Arikayce™
Number analyzed (Participants) | 49
Log 10 CFU/mL
  Baseline | 6.289 (2.8587)
  Day 14: number analyzed (Participants) | 37
  Day 14 | -1.196 (2.0736)
  Day 28: number analyzed (Participants) | 43
  Day 28 | -0.416 (1.8584)
  Day 85: number analyzed (Participants) | 40
  Day 85 | 0.154 (2.4433)
  Day 98: number analyzed (Participants) | 39
  Day 98 | -0.623 (1.9127)
  Day 112: number analyzed (Participants) | 38
  Day 112 | -0.781 (1.1625)
  Day 140: number analyzed (Participants) | 2
  Day 140 | -0.266 (0.2871)
  Day 169: number analyzed (Participants) | 33
  Day 169 | -0.144 (1.2470)
  Day 182: number analyzed (Participants) | 30
  Day 182 | -1.087 (1.9582)
  Day 196: number analyzed (Participants) | 31
  Day 196 | -0.599 (1.3450)
  Day 253: number analyzed (Participants) | 31
  Day 253 | 0.213 (1.4059)
  Day 266: number analyzed (Participants) | 33
  Day 266 | -0.991 (2.5040)
  Day 280: number analyzed (Participants) | 33
  Day 280 | -0.702 (1.7419)
  Day 337: number analyzed (Participants) | 35
  Day 337 | 0.375 (1.9924)
  Day 350: number analyzed (Participants) | 36
  Day 350 | -0.311 (1.6342)
  Day 364: number analyzed (Participants) | 37
  Day 364 | -0.107 (1.8027)
  Day 421: number analyzed (Participants) | 34
  Day 421 | 0.494 (2.0058)
  Day 434: number analyzed (Participants) | 34
  Day 434 | 0.111 (1.9098)
  Day 448: number analyzed (Participants) | 34
  Day 448 | 0.034 (2.0020)

4. Secondary Outcome: Antipseudomonal Rescue Therapy - Duration of Therapy
Description: The duration of IV and all systemic or inhaled antipseudomonal rescue therapy is presented for the overall safety population and by treatment received.
Time Frame: 18 Months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 560 mg Arikayce™
Number analyzed (Participants) | 49
days | 39.7 (44.57)

5. Secondary Outcome: Antipseudomonal Rescue Therapy - Time to Therapy
Description: The time to IV and all systemic or inhaled antipseudomonal rescue therapy is presented for the overall safety population and by treatment received.
Time Frame: 18 Months
Measure: Number; unit: percentage % participants
Arm/Group | 560 mg Arikayce™
Number analyzed (Participants) | 49
percentage % participants
  By Day 85 | 2.0
  By Day 253 | 17.2
  By Day 504 | 32.9

6. Secondary Outcome: Analysis of Cystic Fibrosis Questionnaire - Revised (CFQ-R) for Absolute Change in Score
Description: A summary of absolute change from baseline in the CFQ-R scales at each on-treatment assessment between Day 14 and Day 448 is presented for all patients and by main study treatment group for the safety population. CFQ-R is a disease specific instrument designed to measure impact on overall health, daily life, perceived well-being and symptoms on a scale from 0 to 100 points. Higher values represent a more favorable outcome.
Time Frame: Days 14, 28, 85, 98, 112, 169, 182,196, 253, 266, 280, 337, 350, 364, 421, 434, and 448
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage %
Arm/Group | 560 mg Arikayce™
Number analyzed (Participants) | 49
percentage %
  Day 14: number analyzed (Participants) | 48
  Day 14 | 7.616 (14.1662)
  Day 28: number analyzed (Participants) | 46
  Day 28 | 11.486 (14.9347)
  Day 85: number analyzed (Participants) | 44
  Day 85 | 9.697 (12.9834)
  Day 98: number analyzed (Participants) | 45
  Day 98 | 11.235 (14.5552)
  Day 112: number analyzed (Participants) | 44
  Day 112 | 11.768 (13.9321)
  Day 169: number analyzed (Participants) | 42
  Day 169 | 5.159 (13.6851)
  Day 182: number analyzed (Participants) | 42
  Day 182 | 9.233 (16.3635)
  Day 196: number analyzed (Participants) | 41
  Day 196 | 9.404 (12.4334)
  Day 253: number analyzed (Participants) | 40
  Day 253 | 7.097 (13.7509)
  Day 266: number analyzed (Participants) | 41
  Day 266 | 10.041 (14.5240)
  Day 280: number analyzed (Participants) | 40
  Day 280 | 6.111 (11.3611)
  Day 337: number analyzed (Participants) | 39
  Day 337 | 9.017 (13.8786)
  Day 350: number analyzed (Participants) | 39
  Day 350 | 12.108 (13.8668)
  Day 364: number analyzed (Participants) | 40
  Day 364 | 11.875 (12.9679)
  Day 421: number analyzed (Participants) | 39
  Day 421 | 11.895 (14.1632)
  Day 434: number analyzed (Participants) | 39
  Day 434 | 13.718 (13.1377)
  Day 448: number analyzed (Participants) | 39
  Day 448 | 13.120 (14.0144)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | 560 mg Arikayce™
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 15/49
Other Adverse Events (participants affected / at risk) | 29/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 560 mg Arikayce™ (N=49)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 11 (17)
Endocarditis (Infections and infestations) | 1 (2)
Appendicitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Endoscopy (Investigations) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1)
Testicular appendage torsion (Reproductive system and breast disorders) | 1 (1)
Drug therapy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 560 mg Arikayce™ (N=49)
Nasopharyngitis (Infections and infestations) | 14 (26)
Rhinitis (Infections and infestations) | 11 (19)
Influenza (Infections and infestations) | 6 (7)
Respiratory tract infection viral (Infections and infestations) | 5 (12)
Pharyngitis (Infections and infestations) | 5 (5)
Sinusitis (Infections and infestations) | 4 (4)
Bronchitis (Infections and infestations) | 3 (6)
Viral rhinitis (Infections and infestations) | 3 (4)
Viral infection (Infections and infestations) | 3 (3)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 24 (67)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (33)
Haemopytsis (Respiratory, thoracic and mediastinal disorders) | 12 (20)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 (14)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 (13)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 4 (5)
Abdominal Pain upper (Gastrointestinal disorders) | 3 (4)
Pyrexia (General disorders) | 5 (7)
Blood alkaline phosphatase increased (Investigations) | 3 (4)
Headache (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the signed Investigator Agreement in the study protocol and protocol amendments, the PI agreed "not to originate or use the name of Insmed Incorporated, or study drug code in any publicity, news release, or other public announcement, written or oral, whether to the public, press, or otherwise, relating to this protocol, to any amendment to the protocol, or to the performance of this protocol, without the prior written consent of Insmed Incorporated."